CLINICAL TRIAL: NCT06570174
Title: Oral Protein Supplements Might Improve Nutritional Status and Quality of Life in Elderly Patients After Standard Pancreatic Resection
Brief Title: Oral Protein Supplements for Nutritional and Quality of Life Improvement After Pancreatic Resection in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 4-2020-0552
Record Dates: First submitted 2024-08-18; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer; Cholangiocarcinoma; Intraductal Papillary Mucinous Neoplasm; Neuroendocrine Tumor; Solid Pseudopapillary Tumor
MeSH Terms: conditions — Pancreatic Neoplasms; Cholangiocarcinoma; Neuroendocrine Tumors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein Supplement group (Experimental): This group received a daily oral protein supplement providing 18g of protein. The supplement was administered postoperatively and continued throughout the study period to evaluate its impact on nutritional status, quality of life, muscle mass, muscle strength, and gait speed.
  Interventions: Dietary Supplement: oral protein supplements
- Placebo group (Placebo Comparator): This group received a placebo that contained carbohydrates instead of protein. The placebo was identical in appearance and taste to the protein supplement, ensuring the double-blind nature of the study. This arm was used to compare the effects of the protein supplement on the same outcomes.
  Interventions: Genetic: placebo

INTERVENTIONS:
Dietary Supplement: oral protein supplements — Participants in this group received an oral protein supplement providing 18g of protein per day. The supplement was administered postoperatively and continued throughout the study period. The goal was to assess the impact of protein supplementation on protein intake, nutritional status, quality of life, muscle mass, muscle strength, and 10-meter gait speed. These outcomes were measured at three specific time points: before surgery, at discharge, and during the outpatient visit.
  Arms: Protein Supplement group
Genetic: placebo — Participants in this group received a placebo supplement containing carbohydrates instead of protein, which was identical in appearance and taste to the protein supplement to maintain the study's double-blind design. The placebo was administered postoperatively and continued throughout the study period. The aim was to serve as a control to evaluate the effects of the protein supplement on outcomes including nutrient intake, nutritional status, quality of life, muscle mass, muscle strength, and 10-meter gait speed, measured at three key time points: before surgery, at discharge, and during the outpatient visit.
  Arms: Placebo group

SUMMARY:
This study investigates the effects of oral protein supplements on the nutritional status and quality of life in elderly patients following standard pancreatic resection. The research aims to determine whether these supplements can improve protein intake and contribute to better skeletal muscle mass, which is critical for recovery and overall health. The study hypothesizes that higher compliance with protein supplementation will be positively correlated with increased protein intake and improved muscle mass index, potentially leading to enhanced postoperative outcomes in this patient population.

DETAILED DESCRIPTION:
This study was a randomized, double-blind, placebo-controlled clinical trial conducted to assess the effects of oral protein supplements on nutritional status and quality of life in elderly patients following pancreaticobiliary surgery. The study included elderly patients aged 65 years or older who underwent surgery for pancreaticobiliary cancer. The trial was conducted between January 7, 2021, and July 18, 2022.

A total of 60 patients were initially enrolled, but after 19 dropouts, the final analysis was based on 41 patients (18 in the placebo group and 23 in the experimental group). The experimental group received protein supplements providing 18g of protein per day, while the control group received a placebo containing carbohydrates instead of protein.

Key outcomes such as nutrient intake, nutritional status, quality of life, muscle mass, muscle strength, and 10-meter gait speed were measured at three time points: before surgery, at discharge, and during an outpatient visit. The data were analyzed using a Linear Mixed-Effects Model to evaluate the effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years or older who were diagnosed with and underwent surgery for one of the following cancers:

  1. pancreatic cancer
  2. cholangiocarcinoma
  3. intraductal papillary mucinous neoplasm
  4. neuroendocrine tumor
  5. solid pseudopapillary tumor.

Exclusion Criteria:

* Patients were excluded from the study if they met any of the following criteria:

  1. Patients who were assessed as severely malnourished before surgery (PG-SGA grade C);
  2. Patients with an estimated glomerular filtration rate (eGFR) of less than 60 mL/min, or those diagnosed with chronic kidney disease and a history of related treatment;
  3. Patients with a body mass index (BMI) of 30 kg/m² or higher;
  4. Patients with ascites or edema severe enough to affect weight evaluation;
  5. Patients whose bioelectrical impedance analysis (BIA) could not be measured due to the use of pacemakers or implants;
  6. Patients whom the researcher deemed unable to participate in the study for psychological or cognitive reasons;
  7. Patients who did not provide consent for participation in this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Muscle mass | 1. The day before surgery (pre-OP), 2. Within 24 hours before the scheduled discharge date (DC; approximately 5 to 7 days postoperatively), 3. At the first outpatient visit following surgery (OPD; approximately 6 weeks postoperatively)."
  Muscle mass was measured using the InBody S10 (InBody®, Seoul, Korea) device, which employs the Bioelectrical Impedance Analysis (BIA) method. Body Cell Mass (BCM), Phase Angle, and Skeletal Muscle Mass Index (SMI) were used for analysis. The SMI was calculated by dividing the appendicular skeletal muscle mass (ASM), which is the sum of the muscle mass of the limbs excluding the trunk, by the square of the height in meters [SMI = ASM/height²].
nutritional status | 1. The day before surgery (pre-OP), 2. Within 24 hours before the scheduled discharge date (DC; approximately 5 to 7 days postoperatively), 3. At the first outpatient visit following surgery (OPD; approximately 6 weeks postoperatively)."
  Nutritional status was assessed using the Patient-Generated Subjective Global Assessment (PG-SGA). This tool involves patient-reported changes in weight, food intake, symptoms affecting intake, and activity level. A dietitian then evaluates factors like diagnosis, metabolic stress, body fat, muscle mass, and edema to classify the patient's nutritional status as well-nourished (Grade A), moderately malnourished (Grade B), or severely malnourished (Grade C).

SECONDARY OUTCOMES:
Intake | 1. The day before surgery (pre-OP), 2. Within 24 hours before the scheduled discharge date (DC; approximately 5 to 7 days postoperatively), 3. At the first outpatient visit following surgery (OPD; approximately 6 weeks postoperatively)."
  Usual intake before surgery was investigated using the 24-hour recall method. During the hospitalization period, the patients' daily intake was recorded using the self-developed "meal intake during hospitalization" survey. The patients were asked to write a "meal journal" and bring it with them at the time of their first outpatient visit. The patients' nutrient intake was analyzed using the "CAN-Pro 5.0(Web ver.) (Korean Nutrition Society, Seoul, Korea)" program.
QoL | 1. The day before surgery (pre-OP), 2. Within 24 hours before the scheduled discharge date (DC; approximately 5 to 7 days postoperatively), 3. At the first outpatient visit following surgery (OPD; approximately 6 weeks postoperatively)."
  The patients' quality of life was assessed using the "European Organization for Research and Treatment in Cancer 30 (EORTC QLQ-C30)" questionnaire, which is a questionnaire designed to evaluate the quality of life of cancer patients. The final score was calculated by adding the scores for the last two questions out of 30 evaluation questions on the subjects' overall quality of life. The higher the quality of life (QoL) score, the better the quality of life.
Walking Speed(Indicators Related to Sarcopenia) | 1. The day before surgery (pre-OP), 2. Within 24 hours before the scheduled discharge date (DC; approximately 5 to 7 days postoperatively), 3. At the first outpatient visit following surgery (OPD; approximately 6 weeks postoperatively)."
  The time it took for the patients to walk 10 meters on a straight and flat surface was measured. Gait speed was measured in the hallway of the hospital ward during hospitalization and in the corridor of the clinic during outpatient visits. The patients were in structed to walk at their usual pace.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No